CLINICAL TRIAL: NCT00205101
Title: Clinical Outcome Study of the Triad Allograft for Posterior Lumbar Fusion
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: NuVasive (Industry)
Responsible Party: Sponsor
Other Study IDs: HSC# 2004-0235
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Pain; Stenosis; Spondylolisthesis
Keywords: Transforaminal lumbar interbody fusion; Posterior lumbar interbody fusion; Isthmic spondylolisthesis, degenerative spondylolisthesis; Pseudoarthritis; Severe Foraminal Stenosis
MeSH Terms: conditions — Pain; Constriction, Pathologic; Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- 1: Triad allograft
- 2: other anterior lumbar interbody fusion (ALIF)
- 3: transforaminal lumbar interbody fusion (TLIF)
- 4: posterior lumbar interbody fusion (PLIF)

SUMMARY:
The purpose of the study is to prospectively measure pain, function, and patient satisfaction in 70 consecutive patients treated by lumbar fusion using the Triad allograft. Results of the Triad allograft will be compared to those of other anterior lumbar interbody fusion (ALIF), transforaminal lumbar interbody fusion (TLIF), and posterior lumbar interbody fusion (PLIF) surgeries. Patient participation is based on the physician determination that the patient requires one of these surgeries. Participants will be evaluated pre-operatively and post-operatively at 3, 6, 12,and 24 month intervals. Clinic procedures will be related to standard of care except for the completion of several study questionnaires:

1. Back Pain Questionnaire;
2. Oswestry Disability Index Questionnaire;
3. Short Form-36 (SF-36) Survey;
4. Visual Analog Pain Scale (VAS); and
5. The Modems Patient Satisfaction Survey.

Outcome Measurements:

1. The patient's pain is scored by a VAS normalized to 100;
2. Patient function is based on Oswestry scores;
3. General health is assessed by SF-36 completion; and
4. Overall patient satisfaction will be determined by the completion of the Modems.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary consent for an observational study
2. One of the following diagnoses:

   * isthmic spondylolisthesis,
   * degenerative spondylolisthesis,
   * pseudoarthritis,
   * severe foraminal stenosis, and
   * prior failed discectomies
3. Single, two, or three level fusions
4. Patients require treatment by TLIF or PLIF posterior fusion as determined by surgeon. Pedicle screw instrumentation will be placed in all cases.

Exclusion Criteria:

1. Infection at operative site
2. Severe osteoporosis
3. Inability to return for follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 70 consecutive patients treated by lumbar fusion using the Triad allograft
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2004-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Anderson, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Health Spine Clinic, Madison, Wisconsin, United States